CLINICAL TRIAL: NCT02437539
Title: 68Ga-NOTA-AE105. Evaluation of a New Radiotracer Targeting uPAR (Urokinase Plasminogen Activator Receptor), for Positron Emission Tomography Imaging of the Invasive Cancer Phenotype. First in Human
Brief Title: Evaluation of a New Radiotracer (68Ga-NOTA-AE105) for Diagnosing Aggressive Cancer With Positron Emission Tomography
Acronym: uPAR-PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Curasight (Industry)
Responsible Party: Principal Investigator, Dorthe Skovgaard, MD, Phd, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-730; 2014-005522-35 (EudraCT Number)
Record Dates: First submitted 2015-04-28; First posted 2015-05-07 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer; Prostate Cancer; Urinary Bladder Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-NOTA-AE105 PET (Experimental): One injection of 68Ga-NOTA-AE105 (app. 200 MBq) followed by 3 PET/CT scans 10 minutes, 1 hour and 2 hours post injection
  Interventions: Drug: Injection of 68Ga-NOTA-AE105; Device: Positron Emission Tomography scans

INTERVENTIONS:
Drug: Injection of 68Ga-NOTA-AE105 — One injection of 68Ga-NOTA-AE 105
Device: Positron Emission Tomography scans — Following injection of 68Ga-NOTA-AE105 the patients will be PET scanned at 10 minutes, 1 hour and 2 hours post injection

SUMMARY:
The primary objective of the study is to test a new radiotracer called 68Ga-NOTA-AE105 for PET imaging of uPAR (urokinase plasminogen activator receptor). The tracer has the potential of identifying the invasive cancer phenotype, thereby distinguishing between aggressive and less aggressive tumors. This is a first in human study to test the radiotracer in cancer patients. The biodistribution and tumor uptake will be evaluated by repeated PET imaging (10 minutes, 1 hour and 2 hours post injection).

DETAILED DESCRIPTION:
The primary objective of the study is to test a new radiotracer called 68Ga-NOTA-AE105 for PET imaging of uPAR (urokinase plasminogen activator receptor). The tracer has the potential of identifying the invasive cancer phenotype, thereby distinguishing between aggressive and less aggressive tumors. This is a first in human study to test the radiotracer in cancer patients. The biodistribution and tumor uptake will be evaluated by repeated PET scans (10 minutes, 1 and 2 hours post injection). The primary end points are safety, biodistribution and dosimetry of 68Ga-NOTA-AE105. In addition, the quantitative uptake of 68Ga-NOTA-AE105 will be compared to the expression of uPAR measured directly in tumor tissue obtained by surgery or biopsies. The project will be monitored and evaluated in accordance with the principles of Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with cancer of prostate, breast or urinary bladder
2. capable of understanding and giving full informed consent

Exclusion Criteria:

1. pregnancy
2. lactation
3. contraindication for the use of intravenous CT contrast-agencies
4. claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Biodistribution | 2 hours
  The patients will be PET scanned 10 minutes, 1 hour and 2 hours post injection of the radiotracer 68Ga-NOTA-AE105. These timepoints will be used for assessment of biodistribution
Dosimetry | 2 hours
  The patients will be PET scanned 10 minutes, 1 hour and 2 hours post injection of the radiotracer 68Ga-NOTA-AE105. These timepoints will be used for calculation of dosimetry with the use of OLINDA/EXM software (mSv)
Safety | 2 hours
  the patients will be monitored for safety (occurence of adverse events, vital signs, blood test parameters) following injection of the radiotracer 68Ga-NOTA-AE105

SECONDARY OUTCOMES:
Quantitative uptake of the radiotracer in tumor tissue | 2 hours
  The patients will be PET scanned 10 minutes, 1 hour and 2 hours post injection of the radiotracer 68Ga-NOTA-AE105. These timepoints will be used for assessment of tumor uptake

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Skovgaard, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Result] Persson M, Madsen J, Ostergaard S, Jensen MM, Jorgensen JT, Juhl K, Lehmann C, Ploug M, Kjaer A. Quantitative PET of human urokinase-type plasminogen activator receptor with 64Cu-DOTA-AE105: implications for visualizing cancer invasion. J Nucl Med. 2012 Jan;53(1):138-45. doi: 10.2967/jnumed.110.083386. PMID 22213823